CLINICAL TRIAL: NCT04841421
Title: Clinical Study on Positron Emission Tomography (PET) Imaging, Distribution and Pharmacokinetics of 89 Zirconium (Zr)-CD147 in Patients With Solid Tumors
Brief Title: Clinical Study on PET Imaging, Distribution and PK of 89Zr-CD147 in Patients With Solid Tumors
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Principal Investigator, Yue Chen, Director, The Affiliated Hospital Of Southwest Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: STB017
Record Dates: First submitted 2021-02-06; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 89Zr-CD147 1mCi±10% 10mg dose group (Experimental): The activity administered was 1mCi±10% and the mass of radiolabeled CD147 was 10 mg.
  Interventions: Drug: 89Zr-CD147
- 89Zr-CD147 3mCi±10% 10mg dose group (Experimental): The activity administered was 3mCi±10% and the mass of radiolabeled CD147 was 10 mg.
  Interventions: Drug: 89Zr-CD147
- 89Zr-CD147 5mCi±10% 10mg dose group (Experimental): The activity administered was 5mCi±10% and the mass of radiolabeled CD147 was 10 mg.
  Interventions: Drug: 89Zr-CD147

INTERVENTIONS:
Drug: 89Zr-CD147 — The 89Zr-CD147 is a promising positron emission tomography probe and it is possible to select suitable tumor patients with CD147 expression to benefit from anti-CD147 treatment.

SUMMARY:
The primary objective of this study is to observe the distribution of 89Zr-CD147 and radiation dosimetry characteristics in patients with solid tumors. The secondary objective is to observe the pharmacokinetic characteristics of 89Zr-CD147 in patients with solid tumors. This study is a single-center, open-lable study, including 89Zr-CD147 1mCi±10%，89Zr-CD147 3mCi±10% and 89Zr-CD147 5mCi±10% dose group. The trial is expected to last for 2 years from the first patient signing the consent form to the end of the trial.

DETAILED DESCRIPTION:
Antibody based positron emission tomography (immuno-PET) imaging is of increasing importance to visualize and characterize tumor lesions. Additionally, it can be used to identify patients who may benefit from a particular therapy and monitor the therapy outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be between 18 and 70 years old (including 18 and 70 years old), male or female;
2. Patients with advanced solid tumors (stage IV): non-small cell lung cancer (NSCLC); Gastric adenocarcinoma; Colorectal adenocarcinoma, etc ;
3. Patients must have an ECOG performance status of 0-1;
4. Patients must have a life expectancy ≥ 12 weeks;
5. Patients must have adequate organ function:

   White blood cell (WBC) count≥4.0x10^9/L or absolute neutrophil count (ANC) ≥1.5 x 10^9/L, Platelets ≥100 x 10^9/L, Hemoglobin≥ 90g/L ; thrombin time or Activated partial thromboplastin time≤1.5ULN; liver and renal function: Total bilirubin≤1.5ULN (upper limit of normal), Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)≤2.5ULN or ≤5ULN (subjects with liver metastasis), alkaline phosphatase (ALP)≤ 2.5ULN (if there is bone metastasis or liver metastasis ALP≤4.5ULN). Urea (BUN)≤1.5ULN, creatinine≤1.5ULN;
6. Patients must have ≥1 measurable lesion according to RECIST1.1 criteria;
7. For patients who have partners of childbearing potential: Partner and/or patient must use a method of birth control with adequate barrier protection, deemed acceptable by the principle investigator during the study and for 6 months after last study drug administration.;
8. Patients must have the ability to understand and sign an approved ICF.

Exclusion Criteria:

1. There are any of the following conditions, such as brain metastasis (except for asymptomatic primary or metastatic brain tumors that do not need treatment), carcinomatous meningitis, myocardial infarction (within 6 months before enrollment), unstable angina pectoris, or high risk of uncontrollable arrhythmia, coronary artery bypass grafting, cerebrovascular accident (within 6 months before enrollment), congestive heart failure (cardiac function grade III-IV), pulmonary embolism, deep venous thrombosis, Infections that need to be treated with intravenous antibiotics within 2 weeks, and immunosuppressant therapy after organ transplantation;
2. Primary central nervous system tumor;
3. HBV DNA≥1000 copies/ml;
4. HCV-RNA≥1000 copies/ml;
5. People with positive antibodies to HIV or syphilis;
6. Patients with acute or subacute intestinal obstruction, or a history of inflammatory bowel disease;
7. Women who are pregnant, breastfeeding or planning pregnancy;
8. People who are known to be allergic to the study preparation or its auxiliary materials;
9. People with a history of psychotropic substance abuse and inability to get rid of it or mental disorders;
10. Patients who cannot lie for half an hour;
11. Patients who are allergic to any component of the imaging agent or antibody;
12. Patients who cannot accept PET/CT imaging;
13. Situations that other researchers consider unsuitable to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | Day 0-7
  Standardized uptake value of tumor
standardized uptake value ratio (SUVR) | Day 0-7
  The ratio of the standardized uptake value of the tumor or suspected tumor lesion to the standardized uptake value of normal tissue
Radiation dose | Day 0-7
  Radiation dose of whole body and major tissues / organs of subjects after administration

SECONDARY OUTCOMES:
Terminal Half Time (T1/2) | Day 0-7
  Pharmacokinetic parameters
Clearance (CL) | Day 0-7
  Pharmacokinetic parameters
Peak Plasma Concentration (Cmax) | Day 0-7
  Pharmacokinetic parameters
Area under the plasma concentration versus time curve (AUC) | Day 0-7
  Pharmacokinetic parameters
Distribution (dL) | Day 0-7
  Pharmacokinetic parameters

IPD SHARING:
Plan to Share IPD: No